CLINICAL TRIAL: NCT05309668
Title: A Phase I/II, Single-Arm, Open Label Study to Evaluate the Pharmacokinetics, Safety/Tolerability and Efficacy of the Selumetinib Granule Formulation in Children Aged ≥1 to <7 Years With Neurofibromatosis Type 1 (NF1) Related Symptomatic, Inoperable Plexiform Neurofibromas (PN) (SPRINKLE)
Brief Title: Pharmacokinetics, Safety and Efficacy of the Selumetinib Granule Formulation in Children Aged ≥1 to <7 Years With NF1-related Symptomatic, Inoperable PN
Acronym: SPRINKLE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1346C00004; D1346C00004 (Registry Identifier: CTIS (EU)); 2020-005608-20 (EudraCT Number)
Record Dates: First submitted 2021-11-26; First posted 2022-04-04 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — AZD 6244; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selumetinib single arm (Experimental): This study consists of a screening period (up to 28 days), a treatment period (25 cycles) and a long term safety follow-up for participants until they are 5 years old or commence an alternative systemic NF1-PN treatment, whichever is the earlier. Participants may continue treatment with selumetinib throughout the long term safety follow-up as long as they are considered to be receiving clinical benefit in the opinion of their Investigator. A safety follow up assessment will be performed 30 days after the last dose of study intervention for all study participants.
  Interventions: Drug: Selumetinib granule formulation; Drug: Selumetinib capsule formulation

INTERVENTIONS:
Drug: Selumetinib granule formulation — Selumetinib granule formulation will be administered using BSA-based dosing. The granule formulation dose schema to be used in the study will be established in the dose finding phase.
  At enrolment participants must have a BSA within the range 0.40 to 1.09 m2; once participants attain a BSA between 1.10 and 1.29 m2 they will be encouraged to transition to the capsule formulation, if feasible, although all participants must remain on the granule formulation until after they have completed their third cycle of treatment.
Drug: Selumetinib capsule formulation — Selumetinib capsule formulation will be administered using BSA-based dosing. Once participants attain a BSA between 1.10 and 1.29 m2 they will be encouraged to transition to the capsule formulation, if feasible, although all participants must remain on the granule formulation until after they have completed their third cycle of treatment.

SUMMARY:
This study is designed to define a dosing regimen and assess the pharmacokinetics(PK) and safety of the granule formulation; the study will also include descriptive analyses of exploratory efficacy endpoints. The study will inform the benefit risk profile of the granule formulation in children aged ≥ 1 to < 7 years with NF1 related symptomatic, inoperable PN.

DETAILED DESCRIPTION:
This is a Phase I/II, single arm, open-label study in children aged ≥ 1 to < 7 years at study entry (date of ICF signature) with a clinical diagnosis of NF1 related symptomatic, inoperable PN. The study is designed to evaluate the PK, safety and tolerability of selumetinib given as a granule formulation.

Participants will receive selumetinib for 25 cycles (or until they meet discontinuation criteria). Enrolment into the initial dose-finding phase will be stratified by age group:

* Cohort 1: participants aged between ≥ 4 and < 7 years
* Cohort 2: participants aged between ≥ 1 to < 4 years

In addition to the Global Cohorts, 6 Japanese participants in Japan aged between ≥ 1 to < 7 years with NF1 related symptomatic, inoperable PN will be enrolled into the Japan Cohort.

After completion of at least one cycle (28 days) of dosing in 3 evaluable participants in Cohort 1, Safety Review Committee(SRC) will review the emerging safety and PK data. Providing the single dose PK exposure is within the acceptable range and there are no safety concerns as determined by SRC then dosing in Cohort 2 will be initiated and additional participants will be dosed in Cohort 1. If the PK exposure is not within the acceptable range, the dose schema may be adjusted to ensure that selumetinib exposure is within the range observed in the SPRINT study; PK will be assessed against acceptance criteria in an additional 3 evaluable cohort 1 participants who received the adjusted dose. Cohort 2 will be initiated once the selumetinib granule formulation dose schema is identified for Cohort 1. The physiologically-based PK model will be updated, if required, based on emerging PK data.

Additional SRC reviews will be held for each of the cohorts following at least one cycle of dosing in approximately 6 evaluable participants and again in approximately 10 evaluable participants. The SRC will evaluate the PK, safety and tolerability of the granule formulation for that dose schema. The Japan Cohort will not participate in the dose-finding phase.

Participants who are aged ≥ 5 years at the end of 25 cycles of selumetinib will be considered to have completed the study for data analysis purposes. Participants who terminate treatment prior to Cycle 25 will be followed up to collect MRIs performed as standard of care and details of NF1-PN treatment information until the time when they would have completed 25 cycles of treatment, or they commence an alternative systemic NF1-PN treatment, whichever is the earliest. Any participant who is aged < 5 years after 25 cycles of selumetinib (or when they terminate treatment with selumetinib) will enter a safety follow-up phase. Participation in the safety follow-up will continue until they reach the age of 5 years or commence an alternative systemic NF1-PN treatment, whichever is the earlier. Participants can continue to receive selumetinib (capsule or sprinkle capsule) during the safety follow-up as long as they are considered to be receiving benefit in the opinion of their Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged ≥ 1 to < 7 years of age at the time their legally authorised representative (parent or guardian) signs the informed consent.
2. All study participants must be diagnosed with NF1 with symptomatic inoperable PN as defined in protocol.
3. Participants must have at least one measurable PN, defined as a PN of at least 3 cm measured in one dimension, which can be seen on at least 3 imaging slices and have a reasonably well-defined contour. Participants who have undergone surgery for resection of a PN are eligible provided the PN was incompletely resected and is measurable. The target PN will be defined as the clinically most relevant PN, which is symptomatic, inoperable and measurable by volumetric MRI analysis.
4. Performance status: Participants must have a Lansky performance of ≥ 70 except in participants who are wheelchair bound or have limited mobility secondary to a need for mechanical breathing support (such as an airway PN requiring tracheostomy or continuous positive airway pressure) who must have a Lansky performance of ≥ 40.
5. Participants must have a BSA ≥ 0.4 and ≤ 1.09 m2 at study entry (date of ICF signature).
6. Mandatory provision of consent for the study signed and dated by a participant's legally authorised representative (parent or guardian) along with the paediatric assent form, if applicable.

Exclusion Criteria:

1. Participants with confirmed or suspected malignant glioma or MPNST. Participants with low grade glioma (including optic glioma) not requiring systemic therapy are permitted.
2. History of malignancy except for malignancy treatment with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk of recurrence.
3. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of selumetinib.
4. A life-threatening illness, medical condition, organ system dysfunction or laboratory finding which, in the Investigator's opinion, could compromise the participant's safety, interfere with the absorption or metabolism of selumetinib, or put the study outcomes at undue risk.
5. Participants with clinically significant cardiovascular disease as defined in the protocol.
6. Liver function tests: Bilirubin > 1.5 × the ULN for age with the exception of those with Gilbert syndrome (≥ 3 × ULN) or AST/ALT > 2 × ULN.
7. Renal Function: Creatinine clearance or radioisotope glomerular filtration rate < 60 mL/min/1.73 m2 or Serum creatinine > 0.8 mg/dL (for participants aged ≥ 1 to < 4 years) or > 1.0 mg/dL (for participants aged ≥ 4 years).
8. Participants with ophthalmological findings/condition as listed in the protocol.
9. Have any unresolved chronic toxicity with CTCAE Grade ≥ 2 which are associated with previous therapy for NF1-PN (except hair changes such as alopecia or hair lightening)
10. Participants who have previously been treated with a MEKi (including selumetinib) and have had disease progression, or due to toxicity have either discontinued treatment and/or required a dose reduction.
11. Have inadequate haematological function defined as: An absolute neutrophil count < 1500/μL or Haemoglobin < 9g/dL or Platelets <100,000/μL or Have had a transfusion (of red cells or other blood derived products) within the 28 days prior to study entry (date of ICF signature).
12. Have received or are receiving an IMP or other systemic NF1-PN target treatment (including MEKi) within 4 weeks prior to the first dose of study intervention, or within a period during which the IMP or systemic PN target treatment has not been cleared from the body (eg, a period of 5 'half-lives'), whichever is longer.
13. Has received radiotherapy in the 6 weeks prior to start of study intervention or any prior radiotherapy directed at the target or non-target PN.
14. Receiving herbal supplements or medications known to be strong or moderate inhibitors of the CYP3A4 and CYP2C19 enzymes or inducers of the CYP3A4 enzyme unless such products can be safely discontinued at least 14 days or 5 half-lives (whichever is longer) before the first dose of study medication.
15. Inability to undergo MRI and/or contraindication for MRI examinations. Prosthesis or orthopaedic or dental braces that would interfere with volumetric analysis of target PN on MRI.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-04-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study physician Study physician, MD, Study Director — AstraZeneca
Locations (15):
- United States (4):
  - Research Site, Akron, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
- Germany (3):
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Tübingen
- Italy (2):
  - Research Site, Milan
  - Research Site, Rome
- Japan (2):
  - Research Site, Nagoya
  - Research Site, Setagaya City
- Research Site, Rotterdam, Netherlands
- Research Site, Moscow, Russia
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Hernaiz Driever P, Kordes UR, Brecht IB, Saletti V, Fisher MJ, Doughton G, Arefayene M, Rigazio A, Lluch N, Llorente N, Diede SJ, Salvador H. Pharmacokinetics and Safety of Selumetinib Granule Formulation in Children With Symptomatic, Inoperable Neurofibromatosis Type 1-Related Plexiform Neurofibromas (SPRINKLE; phase I/II). J Clin Oncol. 2026 Jan 27:JCO2501447. doi: 10.1200/JCO-25-01447. Online ahead of print. PMID 41592259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is active, not recruiting and conducted in 7 countries with 39 patients who gave informed consent on or prior to 15 January 2024. Results are reported for the study at data cut-off 1 (DCO1) 08 April 2024.
Pre-assignment Details: Eligible patients aged >= 1 to < 7 years at the time of informed consent with a diagnosis of NF1 with symptomatic inoperable PN fall into one of three cohorts: Global Cohort 1 (>=4 to <7 years), Global Cohort 2 (>=1 to <4 years), or Japan Cohort (>=1 to <7 years).
Groups:
- Global Cohort 1: Global Cohort 1 (>=4 to <7 years)
- Global Cohort 2: Global Cohort 2 (>=1 to <4 years)
- Japan Cohort: Japan Cohort (>=1 to <7 years)
Period: Overall Study
Arm/Group | Global Cohort 1 | Global Cohort 2 | Japan Cohort
Started | 15 | 17 | 4
Completed | 1 | 0 | 0
Not Completed | 14 | 17 | 4
Not completed — Ongoing at data cut-off | 14 | 17 | 4

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on all patients in the who received selumetinib (safety analysis set).
Groups:
- Total: Total of all reporting groups
Arm/Group | Global Cohort 1 | Global Cohort 2 | Japan Cohort | Total
Number analyzed (Participants) | 15 | 17 | 4 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.08 (1.101) | 2.49 (0.819) | 4.43 (2.300) | 3.78 (1.681)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 2 | 14
  Male | 10 | 10 | 2 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 13 | 15 | 4 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 4 | 5
  Black or African American | 0 | 1 | 0 | 1
  White | 9 | 13 | 0 | 22
  Other | 2 | 2 | 0 | 4
  Not Reported | 3 | 1 | 0 | 4
Country [Count of Participants; unit: Participants]
  Germany | 5 | 4 | 0 | 9
  Italy | 3 | 6 | 0 | 9
  Japan | 0 | 0 | 4 | 4
  Russian Federation (the) | 2 | 0 | 0 | 2
  Spain | 4 | 4 | 0 | 8
  United States of America (the) | 1 | 3 | 0 | 4
BSA [Mean (Standard Deviation); unit: m2] | 0.771 (0.1073) | 0.558 (0.0603) | 0.605 (0.1234) | 0.652 (0.1349)
Body surface area group (m2) [Count of Participants; unit: Participants]
  >=0.40 to <0.50 | 0 | 1 | 1 | 2
  >=0.50 to <0.60 | 0 | 11 | 0 | 11
  >=0.60 to <0.70 | 3 | 5 | 3 | 11
  >=0.70 to <0.90 | 10 | 0 | 0 | 10
  >=0.90 to <1.10 | 2 | 0 | 0 | 2
  >=1.10 to <=1.29 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Selumetinib AUC0-12 Derived After Single Dose Administration
Description: To determine the pharmacokinetics of selumetinib after administration of the selumetinib granule formulation
Time Frame: Pre-dose and 1, 2, 3, 4, 6, 8 and 10-12 hours after selumetinib single dose on the first day of study treatment (Cycle 1 Day 1) (each cycle is 28 days)
Population: Pharmacokinetic analysis set was used for analysis. Japan Cohort was not considered for the primary endpoint analysis. Some records were excluded for given visits and analytes due to missing concentration data, issues taking the medication and usage of prohibited medications.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Groups:
- Total in Global: Global Cohorts (>=1 to <7 years)
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global
Number analyzed (Participants) | 13 | 15 | 28
h*ng/mL | 1902 [1647 to 2197] | 1699 [1436 to 2009] | 1790 [1609 to 1993]

2. Primary Outcome: Adverse Events Graded by CTCAE Ver 5.0
Description: To assess the safety and tolerability of the selumetinib granule formulation.
Time Frame: from screening until 30 days after last dose
Reporting Status: Not Posted, anticipated posting 2027-11

3. Secondary Outcome: Palatability Using the Parent-reported Observer Palatability Questionnaire
Description: To assess the palatability of the selumetinib granule formulation
Time Frame: Twice daily (morning and evening), from the first day of study treatment (Cycle 1 Day 1) for one week, from Cycle 7 Day 1 for one week (each cycle is 28 days)
Reporting Status: Not Posted, anticipated posting 2027-11

4. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib AUC0-12 Derived After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose and 1, 2, 3, 4, 6, 8, 10-12 and 18-24 hours after selumetinib single dose on the first day of study treatment (Cycle 1 Day 1). Pre-dose, 1, 2, 3, 4, 6, 8, and 10-12 hours post-dose on Cycle 2 Day 1 (each cycle is 28 days)
Population: Pharmacokinetic analysis set was used for analysis. Some records were excluded for given visits and analytes due to missing concentration data, issues taking the medication and usage of prohibited medications.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
h*ng/mL
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 1902 (24.19) | 1699 (31.02) | 1790 (28.15) | 1526 (25.09)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 13 | 26 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 156.1 (25.76) | 134.0 (34.21) | 144.6 (30.69) | 118.1 (19.56)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 3095 (47.81) | 2114 (49.23) | 2575 (52.23) | 1952 (32.08)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 14 | 14 | 28 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 192.9 (33.37) | 135.9 (33.82) | 161.9 (37.97) | 143.3 (14.64)

5. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib Cmax Derived After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
ng/mL
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 551.1 (44.21) | 464.7 (54.05) | 503.0 (49.58) | 618.4 (76.36)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 40.53 (45.76) | 32.73 (52.62) | 36.14 (49.99) | 43.11 (54.06)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 843.4 (42.69) | 502.6 (58.59) | 656.9 (58.01) | 644.2 (23.68)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 47.53 (38.92) | 29.12 (47.81) | 37.52 (50.63) | 43.20 (19.56)

6. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib AUC0-6 Derived After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose and 1, 2, 3, 4 and 6 hours after selumetinib single dose on the first day of study treatment (Cycle 1 Day 1). Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Cycle 2 Day 1 (each cycle is 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
h*ng/mL
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 1516 (30.42) | 1352 (37.13) | 1426 (34.05) | 1303 (32.65)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 118.3 (31.40) | 99.73 (36.98) | 108.0 (35.04) | 96.22 (28.26)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 2412 (43.55) | 1672 (48.14) | 2021 (49.40) | 1630 (31.40)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 145.6 (31.30) | 102.4 (35.17) | 122.8 (37.71) | 113.0 (14.43)

7. Secondary Outcome: Objective Response Rate
Description: To evaluate the efficacy of the selumetinib granule formulation by assessment of Objective Response Rate
Time Frame: At screening, at week 17 (Cycle5 Day1), week 33 (Cycle9 Day1), week 49 (Cycle13 Day1), week 73 (Cycle19 Day1) and week 97 (Cycle25 Day1), end of treatment (each cycle is 28 days)
Reporting Status: Not Posted, anticipated posting 2027-11

8. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib AUClast Derived After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
h*ng/mL
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 2208 (24.81) | 1932 (29.59) | 2055 (27.85) | 1709 (20.33)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 167.7 (32.98) | 129.7 (38.46) | 146.2 (37.93) | 113.1 (21.03)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 2919 (48.28) | 2031 (49.45) | 2450 (52.12) | 1887 (32.22)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 183.4 (34.54) | 128.9 (34.30) | 154.7 (38.80) | 137.2 (14.86)

9. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib Tmax Derived After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
h
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 1.83 [0.83 to 2.98] | 2.00 [1.00 to 3.88] | 1.97 [0.83 to 3.88] | 2.47 [1.02 to 2.95]
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 1.83 [0.83 to 2.98] | 2.02 [1.00 to 5.87] | 2.00 [0.83 to 5.87] | 2.47 [1.02 to 2.95]
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 2.00 [0.92 to 4.07] | 1.97 [0.92 to 4.05] | 2.00 [0.92 to 4.07] | 1.05 [0.97 to 2.00]
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 2.00 [0.92 to 4.07] | 2.01 [0.92 to 4.05] | 2.00 [0.92 to 4.07] | 1.56 [0.98 to 2.00]

10. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib Tlast Derived After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
h
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 23.10 [21.58 to 24.00] | 23.25 [22.17 to 24.00] | 23.20 [21.58 to 24.00] | 22.43 [21.30 to 22.90]
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 10.12 [10.00 to 24.00] | 10.02 [7.65 to 22.67] | 10.03 [7.65 to 24.00] | 10.23 [7.67 to 10.33]
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 10.00 [8.03 to 12.00] | 10.00 [9.58 to 12.00] | 10.00 [8.03 to 12.00] | 10.23 [10.17 to 10.32]
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 10.00 [8.03 to 12.00] | 10.00 [9.58 to 12.00] | 10.00 [8.03 to 12.00] | 10.23 [10.17 to 10.32]

11. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib AUC0-24 Derived After Single Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose and 1, 2, 3, 4, 6, 8, 10-12 and 18-24 hours after selumetinib single dose on the first day of study treatment (Cycle 1 Day 1) (each cycle is 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 13 | 15 | 28 | 3
h*ng/mL
  Cycle 1 Day 1: Selumetinib | 2222 (24.72) | 1942 (29.73) | 2067 (27.91) | 1568 (7.648)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 13 | 28 | 3
  Cycle 1 Day 1: N-desmethyl selumetinib | 182.4 (27.93) | 148.3 (37.04) | 164.5 (33.92) | 129.8 (13.54)

12. Secondary Outcome: Selumetinib CL/F Derived After Single Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 11
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 12 | 15 | 27 | 3
L/h | 8.411 (19.66) | 6.167 (36.79) | 7.079 (33.95) | 8.757 (2.452)

13. Secondary Outcome: Selumetinib Vz/F Derived After Single Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 11
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 12 | 15 | 27 | 3
L | 91.63 (33.64) | 64.33 (44.81) | 75.28 (43.86) | 107.2 (50.91)

14. Secondary Outcome: Selumetinib t1/2λz Derived After Single Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 11
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 12 | 15 | 27 | 3
h | 7.551 (41.21) | 7.230 (58.00) | 7.371 (49.98) | 8.486 (49.40)

15. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib Rac Cmax Derived After Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, and 10-12 hours post-dose on Cycle 2 Day 1 (each cycle is 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
Ratio
  Cycle 2 Day 1, Selumetinib: number analyzed (Participants) | 15 | 13 | 28 | 4
  Cycle 2 Day 1, Selumetinib | 1.508 (56.59) | 1.104 (92.61) | 1.304 (74.80) | 1.042 (84.39)
  Cycle 2 Day 1, N-desmethyl selumetinib: number analyzed (Participants) | 15 | 13 | 28 | 4
  Cycle 2 Day 1, N-desmethyl selumetinib | 1.142 (61.34) | 0.8837 (76.53) | 1.014 (68.79) | 1.002 (46.75)

16. Secondary Outcome: Selumetinib and N-desmethyl Selumetinib RacAUC0-12 Derived After Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, and 10-12 hours post-dose on Cycle 2 Day 1 (each cycle is 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
Ratio
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 14 | 13 | 27 | 4
  Cycle 2 Day 1: Selumetinib | 1.641 (54.51) | 1.289 (61.20) | 1.461 (58.23) | 1.279 (53.18)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 11 | 24 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 1.221 (35.39) | 1.099 (53.72) | 1.163 (43.69) | 1.213 (23.76)

17. Secondary Outcome: Selumetinib CL/F Derived After Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, and 10-12 hours post-dose on Cycle 2 Day 1 (each cycle is 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 14 | 29 | 4
L/h | 6.166 (50.01) | 6.051 (48.38) | 6.110 (48.25) | 6.943 (26.97)

18. Secondary Outcome: Selumetinib Vss/F Derived After Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, and 10-12 hours post-dose on Cycle 2 Day 1 (each cycle is 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 13 | 28 | 4
L | 33.71 (44.31) | 30.05 (52.48) | 31.96 (47.63) | 31.14 (44.54)

19. Secondary Outcome: Parent-to-metabolite Ratio for AUC0-6, AUC0-12 and AUC0-24 After Single and Multiple Dose Administration.
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose and 1, 2, 3, 4, 6, 8, 10-12 and 18-24 hours after selumetinib single dose on Cycle 1 Day 1. Pre-dose, 1, 2, 3, 4, 6, 8, and 10-12 hours post-dose on Cycle 2 Day 1 (each cycle is 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
Ratio
  Cycle 1 Day 1: MPAUC0-6: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: MPAUC0-6 | 0.07803 (18.27) | 0.07379 (15.50) | 0.07573 (16.76) | 0.07386 (12.37)
  Cycle 1 Day 1: MPAUC0-12: number analyzed (Participants) | 13 | 13 | 26 | 4
  Cycle 1 Day 1: MPAUC0-12 | 0.08204 (17.91) | 0.07722 (17.19) | 0.07960 (17.48) | 0.07742 (14.05)
  Cycle 1 Day 1: MPAUC0-24: number analyzed (Participants) | 13 | 13 | 26 | 3
  Cycle 1 Day 1: MPAUC0-24 | 0.08209 (19.94) | 0.07516 (18.93) | 0.07855 (19.59) | 0.07942 (7.881)
  Cycle 2 Day 1: MPAUC0-6: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: MPAUC0-6 | 0.06036 (29.62) | 0.06123 (26.61) | 0.06078 (27.69) | 0.06934 (20.71)
  Cycle 2 Day 1: MPAUC0-12: number analyzed (Participants) | 14 | 14 | 28 | 4
  Cycle 2 Day 1: MPAUC0-12 | 0.06413 (29.74) | 0.06429 (26.09) | 0.06421 (27.42) | 0.07339 (19.13)

20. Secondary Outcome: Parent to Metabolite Ratio for Cmax After Single and Multiple Dose Administration.
Description: To further evaluate the PK of the granule formulation.
Time Frame: Pre-dose and 1, 2, 3, 4, 6, 8, 10-12, and 18-24 hours post-dose after selumetinib single dose on the first day of treatment (Cycle 1 Day 1). Pre-dose and 1, 2, 3, 4, 6, 8, and 10-12 hours post-dose on Cycle 2 Day 1 (each cycle is 28 days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
Ratio
  Cycle 1 Day 1: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1 | 0.07353 (20.68) | 0.07044 (17.43) | 0.07186 (18.76) | 0.06971 (23.12)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1 | 0.05635 (38.03) | 0.05794 (26.08) | 0.05711 (32.14) | 0.06706 (20.59)

21. Other Pre Specified Outcome: Selumetinib and N-desmethyl Selumetinib BSA Normalised AUC0-6 After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/m2
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
(h*ng/mL)/m2
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 1979 (31.12) | 2446 (40.20) | 2217 (37.31) | 2194 (58.68)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 154.4 (31.96) | 180.5 (38.38) | 167.9 (35.82) | 162.0 (51.74)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 3150 (48.62) | 3038 (48.27) | 3095 (47.53) | 2713 (28.07)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 190.1 (33.01) | 186.0 (34.93) | 188.1 (33.32) | 188.1 (26.55)

22. Other Pre Specified Outcome: Selumetinib and N-desmethyl Selumetinib BSA Normalised AUC0-12 After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/m2
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
(h*ng/mL)/m2
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 2482 (24.78) | 3074 (33.19) | 2784 (31.12) | 2569 (49.75)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 13 | 26 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 203.7 (26.15) | 242.6 (33.67) | 222.3 (30.91) | 198.9 (41.19)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 4041 (54.06) | 3841 (49.45) | 3943 (50.90) | 3249 (27.13)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 14 | 14 | 28 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 247.5 (34.34) | 247.0 (33.49) | 247.2 (33.25) | 238.4 (22.82)

23. Other Pre Specified Outcome: Selumetinib and N-desmethyl Selumetinib BSA Normalised AUClast After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/m2
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
(h*ng/mL)/m2
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 2882 (24.86) | 3496 (31.00) | 3196 (29.58) | 2878 (44.70)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 218.8 (32.79) | 234.8 (37.15) | 227.2 (34.70) | 190.5 (42.43)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 3811 (54.07) | 3690 (49.80) | 3752 (51.02) | 3141 (27.58)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 239.5 (37.31) | 234.2 (34.28) | 236.9 (35.21) | 228.4 (23.68)

24. Other Pre Specified Outcome: Selumetinib and N-desmethyl Selumetinib BSA Normalised Cmax After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/m2
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
(ng/mL)/m2
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 719.2 (47.70) | 840.9 (55.12) | 782.0 (51.47) | 1041 (110.3)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 52.89 (48.40) | 59.23 (52.39) | 56.20 (49.93) | 72.59 (81.41)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 1101 (46.84) | 913.1 (56.39) | 1006 (51.65) | 1072 (32.38)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 62.06 (39.05) | 52.90 (45.74) | 57.46 (42.46) | 71.89 (39.02)

25. Other Pre Specified Outcome: Selumetinib and N-desmethyl Selumetinib Dose Normalised AUC0-6 After Single and Multiple Dose Administration.
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/mg
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
(h*ng/mL)/mg
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 77.91 (30.23) | 104.5 (40.46) | 91.20 (38.73) | 96.12 (55.13)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 6.079 (33.55) | 7.714 (39.05) | 6.906 (38.11) | 7.099 (48.31)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 126.4 (44.74) | 130.7 (47.35) | 128.5 (45.14) | 120.3 (27.94)
  Cycle 2 Day 1: N-desmethyl selumetinib | 7.630 (30.30) | 8.003 (33.93) | 7.808 (31.58) | 8.340 (26.01)

26. Other Pre Specified Outcome: Selumetinib and N-desmethyl Selumetinib Dose Normalised AUC0-12 After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/mg
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
(h*ng/mL)/mg
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 97.73 (23.21) | 131.4 (33.44) | 114.5 (32.58) | 112.6 (46.45)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 13 | 26 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 8.018 (27.48) | 10.31 (34.57) | 9.091 (33.36) | 8.717 (37.98)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 162.2 (50.01) | 165.3 (48.38) | 163.7 (48.25) | 144.0 (26.97)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 14 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 9.935 (30.66) | 10.63 (32.24) | 10.27 (31.05) | 10.57 (22.24)

27. Other Pre Specified Outcome: Selumetinib and N-desmethyl Selumetinib Dose Normalised AUClast After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/mg
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
(h*ng/mL)/mg
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 113.4 (23.10) | 149.4 (31.40) | 131.5 (30.94) | 126.1 (41.51)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 8.615 (33.17) | 10.03 (38.03) | 9.349 (36.09) | 8.347 (39.21)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 152.9 (50.13) | 158.8 (48.72) | 155.7 (48.51) | 139.2 (27.44)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 9.613 (34.31) | 10.08 (33.00) | 9.834 (33.14) | 10.12 (23.11)

28. Other Pre Specified Outcome: Selumetinib and N-desmethyl Selumetinib Dose Normalised Cmax After Single and Multiple Dose Administration
Description: To further evaluate the PK of the granule formulation.
Time Frame: as for outcome 20
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/mg
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort
Number analyzed (Participants) | 15 | 17 | 32 | 4
(ng/mL)/mg
  Cycle 1 Day 1: Selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: Selumetinib | 28.31 (47.51) | 35.94 (55.90) | 32.17 (52.83) | 45.63 (105.5)
  Cycle 1 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 13 | 15 | 28 | 4
  Cycle 1 Day 1: N-desmethyl selumetinib | 2.082 (50.61) | 2.532 (53.47) | 2.312 (52.27) | 3.181 (77.41)
  Cycle 2 Day 1: Selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: Selumetinib | 44.20 (43.64) | 39.29 (55.51) | 41.76 (49.03) | 47.52 (32.01)
  Cycle 2 Day 1: N-desmethyl selumetinib: number analyzed (Participants) | 15 | 14 | 29 | 4
  Cycle 2 Day 1: N-desmethyl selumetinib | 2.491 (38.39) | 2.276 (44.76) | 2.385 (41.03) | 3.187 (38.33)

ADVERSE EVENTS:
Time Frame: All-cause mortality (death due to any cause): from first dose of study medication up to and including the data cut-off 1 analysis (08Apr2024), up to 26 months. Treatment-emergent adverse events: from first dose of study medication up to and including 30 days after the last dose of selumetinib, an average of 12.6 months.
Description: All-cause mortality was reported for all subjects. Adverse events were reported for subjects who received at least one dose of study drug, and includes AEs that start prior to and worsen after treatment or with an onset or worsening date on or after the date of first selumetinib dose up to and including 30 days after the date of last selumetinib dose.
Groups:
- Total in Study: Total in study (>=1 to <7 years)
Arm/Group | Global Cohort 1 | Global Cohort 2 | Total in Global | Japan Cohort | Total in Study
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/32 | 0/4 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/17 | 2/32 | 0/4 | 2/36
Other Adverse Events (participants affected / at risk) | 15/15 | 17/17 | 32/32 | 4/4 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Cohort 1 (N=15) | Global Cohort 2 (N=17) | Total in Global (N=32) | Japan Cohort (N=4) | Total in Study (N=36)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Cohort 1 (N=15) | Global Cohort 2 (N=17) | Total in Global (N=32) | Japan Cohort (N=4) | Total in Study (N=36)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Staring (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (3) | 3 (6) | 0 (0) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 4 (5) | 0 (0) | 4 (5)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (7) | 8 (9) | 0 (0) | 8 (9)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (10) | 8 (9) | 17 (19) | 0 (0) | 17 (19)
Eczema (Skin and subcutaneous tissue disorders) | 6 (7) | 5 (7) | 11 (14) | 3 (3) | 14 (17)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Hair colour changes (Skin and subcutaneous tissue disorders) | 3 (6) | 3 (3) | 6 (9) | 0 (0) | 6 (9)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 3 (4) | 0 (0) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 7 (11) | 13 (17) | 1 (1) | 14 (18)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 8 (8) | 0 (0) | 8 (8)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 5 (5)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (5) | 8 (9) | 12 (14) | 2 (2) | 14 (16)
Fatigue (General disorders) | 4 (4) | 2 (2) | 6 (6) | 0 (0) | 6 (6)
Localised oedema (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (9) | 10 (15) | 16 (24) | 0 (0) | 16 (24)
Swelling face (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anal fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 2 (3)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Cystitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema infectiosum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 5 (7) | 4 (4) | 9 (11) | 0 (0) | 9 (11)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Funguria (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3) | 1 (4) | 3 (7) | 1 (1) | 4 (8)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpangina (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eye oedema (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (6) | 2 (2) | 6 (8) | 0 (0) | 6 (8)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Paronychia (Infections and infestations) | 8 (10) | 7 (14) | 15 (24) | 1 (1) | 16 (25)
Penile infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pustule (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eyelid skin dryness (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 4 (6) | 6 (8) | 0 (0) | 6 (8)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 7 (9) | 11 (14) | 3 (4) | 14 (18)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 3 (4)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 2 (4) | 4 (7) | 0 (0) | 4 (7)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 5 (8) | 5 (6) | 10 (14) | 1 (2) | 11 (16)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 2 (5) | 0 (0) | 2 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2) | 5 (6) | 0 (0) | 5 (6)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Zinc deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Clumsiness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (6) | 0 (0) | 2 (6) | 0 (0) | 2 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The outcome measure "Primary Outcome: Selumetininb AUC0-12₂ Derived After Single Dose Administration" is one of two co-primary endpoints. The second co-primary endpoint - "Adverse Events Graded by CTCAE Version 5.0" - is still ongoing. As a result, the study has not yet reached the Primary Completion Date at the time these results were submitted. Full results, including data for the second co-primary endpoint, will be submitted upon completion of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT05309668/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT05309668/SAP_001.pdf